# 研究方案

项目名称:基于经络-淋巴轴理论的 BMI 分层管理对 妇科肿瘤术后下肢淋巴水肿的干预效果

版本号: V1.0

版本日期: 2025-10-17

主要研究者: 张宏

研究单位: 华中科技大学同济医学院附属同济医院

## 一、研究背景

妇科恶性肿瘤作为严重威胁女性健康的恶性疾病,治疗后下肢淋巴水肿是常见且严重的并发症,严重影响患者生活质量。根据不同的恶性肿瘤病种、不同的随访时间以及诊断方法,下肢淋巴水肿报道的发生率变化范围较大,约为 5%~70%,多数发生在术后 3 年内 [1]。已有研究指出,早期干预在一定程度上有效改善了患者结局 [15]。

综合消肿疗法是治疗淋巴水肿的黄金标准,但患者需要长期且规律地接受费用昂贵的治疗,加上患者本身疾病负担、对疾病的负面态度,在治疗期间容易产生抵抗、担忧及抑郁等不良情绪,导致治疗中断,引发不良预后[2]。现有 CDT 方案多采用 "一刀切" 的模式,未能充分考虑患者个体风险因素的差异,这不仅可能导致医疗护理资源分配不均,还会降低治疗效率,难以满足不同患者的个性化需求 [4]。

在影响妇科肿瘤术后下肢淋巴水肿发生与发展的诸多因素中,身体质量指数已被多项研究证实为强独立危险因素 [1]。随着累积体重每月波动增加,术后下肢淋巴水肿风险也增加,对于术前 BMI>30 并且体重有大幅度波动的患者,会有更高的发生术后下肢淋巴水肿的风险 [3]。临床上需要对此类患者进行密切关注并及早干预,从而更好地进行风险管理 [1,3]。

基于上述临床痛点,本研究提出基于经络一淋巴轴理论的 BMI 分层精准干 预思路,核心依据为 "经络 - 淋巴轴" 理论:现代解剖学证实,足太阴脾经 (三阴交 SP6、阴陵泉 SP9、血海 SP10)、足阳明胃经(足三里 ST36)的体表 循行路径与下肢浅表淋巴管分布重合 [5,6],且穴位刺激可通过激活腓肠神经 CGRP 阳性纤维,增强淋巴管收缩频率(从 3 次 / 分钟提升至 5.2 次 / 分钟),促进淋巴回流 [5,6];同时,BMI 分层可匹配不同代谢状态(如肥胖患者合并慢性炎症,需联合低 GI 饮食调控),旨在降低术后淋巴水肿发生率,兼顾疗效与经济性。

### 二、研究目的

本研究旨在探讨基于经络 - 淋巴轴理论的 BMI 分层干预方案对妇科恶性

肿瘤术后患者 1 个月、3 个月、6 个月下肢淋巴水肿发生率的影响,验证该方案相较于传统 CDT 的精准性与有效性。主要目的:评估该方案对降低淋巴水肿发生率、减轻淋巴水肿相关症状(通过 GCLQ 评分评估)、改善患者生活质量(通过肢体淋巴水肿质量评分评估)以及提高患者自我管理行为的效果。

## 三、研究设计

本研究采用随机对照试验(Randomized Controlled Trial, RCT)设计。从我院妇科肿瘤专科治疗室连续纳入符合标准的妇科恶性肿瘤术后患者。首先,根据 BMI 指数对所有入组患者进行分组:(BMI < 24)、(24 ≤ BMI < 28)、高(BMI ≥ 28)。随后,使用计算机生成的随机数字表,将患者按 1:1 的比例随机分配至实验组或对照组。此过程采用区组随机化以确保组间平衡。四、受试者选择:

纳入标准: (1) 经病理学确诊为妇科恶性肿瘤并行手术治疗(包括淋巴结清扫术)的患者; (2) 年龄 18-75 岁; (3) 意识清楚,能够进行有效沟通,知情同意并自愿参加本研究; (4) 术后生命体征平稳。

排除标准: (1) 术前已存在下肢淋巴水肿、深静脉血栓或淋巴系统疾病; (2) 合并严重心、肝、肾功能不全或其他恶性肿瘤; (3) 存在肢体活动障碍或皮肤疾病影响测量; (4) 伴有认知或精神障碍无法配合研究。

脱落标准: (1) 研究期间肿瘤复发或转移需改变治疗方案; (2) 患者主动要求退出研究; (3) 失访(连续两次无法通过预留联系方式完成随访); (4) 发生严重不良事件,经研究者判断不宜继续参加研究。

# 五、样本量的估算

采用 G\*Power 3.1 软件进行样本量估算。根据预实验或既往文献,设定 α =0.05 (双侧),检验效能(1-β) =0.8,预计效应量(Cohen's d)为 0.8 (大效应量)。主要结局指标为:实验组整体 VS 对照组整体在:预防淋巴水肿效果上的差异。最终将样本量调整至每组 30 例,即按照 BMI 分层的风险等级随机分组,实验组整体 3 0 例,对照组整体 30 例,总共需要纳入 60 例患者。所有数据将采用 SPSS Statistics 25.0 软件进行统计分析。

## 六、研究过程及资料收集方法

#### 6.1 研究工具

- 1. 妇科癌症淋巴水肿问卷(Gynecologic Cancer Lymphedema Questionnaire, GCLQ):该量表包含 20 个症状相关条目,用于筛查和评估淋巴水肿相关症状(如肿胀、疼痛、沉重感等)。总分≥4 分提示存在淋巴水肿,得分越高表示症状负担越重。
- 2. 肢体淋巴水肿生活质量量表(Lymphedema Quality of Life Scale, LYMQOL): 用于评估淋巴水肿对患者生理、心理、社交功能等领域生活质量的影响。得分越低表示生活质量越差。
- 3. 国际淋巴学会分期系统(ISL Staging):
  - Stage 0: 潜伏期或亚临床期,肿胀不明显。
  - Stage I: 凹陷性水肿,抬高患肢可缓解。
  - Stage II: 非凹陷性水肿,组织出现纤维化,抬高患肢不易缓解。
  - Stage III: 象皮肿,患肢极度增粗,伴有皮肤角质化、疣状增生。
- 4. 肢体周径与体积测量:
  - 测量点: 跖趾关节、踝关节(内外踝最窄处), 膝上 10cm, 膝下 10cm。
- 双下肢体积差值比:采用圆台锥截体公式计算下肢体积。单侧肢体体积  $V = \Sigma$  (h /  $12\pi$ ) \* (G  $^2$  +  $C_2$   $^2$  +  $C_4$   $C_2$  ),其中 h 为相邻两测量点间的间隔(10cm),C 和 C 为相邻两测量点的周径。体积差值比 = (患肢体积 健肢体积) / 健肢体积 × 100% 。比值 > 5% 可临床诊断淋巴水肿。

#### 6.2 资料收集方法及过程

- 1. 基线资料收集(术前/T0): 由经过统一培训的研究员在患者入院后、手术前,使用自制的一般资料调查表收集社会人口学资料和临床疾病资料。同时测量并记录双下肢各点周径,计算基线体积。
- 2. 随机分组与干预实施(术后): 患者完成手术后,符合条件者按上述方法进行 BMI 分层和随机分组。实验组按既定方案穴位刺激按摩(指压法),饮食方案护理,对照组接受常规护理。

干预措施:

实验组:接受经络一淋巴轴理论的 BMI 分层精准干预,根据风险层级调整干预强度:

- 1. BMI < 24: 标准健康教育(宣传册 + 口头指导),穴位按摩:三阴交,阴陵泉, 血海(指压法),每穴 3 分钟,每天 3 次,正常饮食,指导自我监测(腿围、沉 重感),常规随访(术后 1、3、6 个月)。
- 2. BMI24-28:增加一对一教育,穴位按摩:三阴交,阴陵泉,血海,(指压法),每穴 5-10 分钟,每天 3 次。饮食方案:控制体重,避免高盐饮食。随访(术后1、3、6 个月)。
- 3. BMI 大于 28 或已有淋巴水肿倾向:穴位按摩:三阴交,阴陵泉,血海,足三里(指压法),每穴 5-10 分钟,每天 3 次。饮食方案:低 GI 高蛋白饮食。建议使用预防性压力袜,建立微信平台进行持续监督与支持,随访(术后 1、3、6个月)。

对照组:接受妇科肿瘤术后常规护理与健康教育,包括发放统一的预防淋巴水肿宣传材料及出院常规指导,并提供门诊随访电话。

所有干预措施由不知晓分组情况的专职护士执行。

3. 随访资料收集: 在术后 1 个月(T1)、3 个月(T2)、6 个月(T3) 对患者进行随访。每次随访时,由另一位不知晓分组情况(盲法评估) 的研究员使用 GCLQ 量表、LYMQOL 量表和卷尺重复测量双下肢周径,并记录国际淋巴水肿分期。 所有数据及时录入电子病例报告表(e-CRF)。

## 七、可能的风险及防范措施

- 1. 隐私泄露风险: 所有收集的资料均采用匿名化编号处理, 电子数据加密存储, 仅限研究团队成员访问。防范措施: 签署保密协议, 使用密码保护的文件和数据库。
- 2. 干预相关风险:实验组患者在进行治疗性运动或手法引流时,可能存在肌肉 拉伤或不适的风险。防范措施:所有干预均在经过培训的专业人员指导下进行, 强度循序渐进。出现任何不适立即停止并评估处理。
- 3. 心理不适风险:谈论疾病并发症可能引起患者焦虑。防范措施:研究人员以同情和鼓励的态度进行沟通,并提供必要的心理支持资源。
- 4. 脱落风险: 因随访时间长,患者可能失访。防范措施:预留多种联系方式,

定期关怀,设置小的激励措施(如免费咨询),合理安排随访时间。

# 八、统计学分析

所有数据采用 SPSS 25.0 软件分析。计量资料若符合正态分布,以均数 ± 标准差 ((x ±s)表示,组间比较采用独立样本 t 检验,组内不同时间点比较采用重复测量方差分析;若非正态分布,以中位数(四分位数间距)[M(IQR)]表示,采用非参数检验(Mann-Whitney U 检验,Wilcoxon 符号秩检验)。计数资料以例数(百分比)[n(%)]表示,采用 x²检验或 Fisher 精确检验。采用广义估计方程(GEE)分析干预措施和时间的交互效应。以 P<0.05 为差异有统计学意义。

## 九、参考文献

- [1] 张佳佳,章孟星,张易,等. 妇科恶性肿瘤患者术后继发性下肢淋巴水肿管理的循证实践 [J]. 护 士 进 修 杂 志 ,2025,40(14):1537-1544. DOI:10.16821/j.cnki.hsjx.2025.14.014.
- [2] 王蕾,朱淑芳,陈翠琴,等. 手法淋巴引流综合消肿疗法在妇科肿瘤淋巴水肿中的临床应 用 [J]. 癌 症 进 展 ,2023,21(3):261-264,268. DOI:10.11877/j.issn.1672-1535.2023.21.03.07.
- [3] 王季, 张意辉, 张丽娟, 等. 体重指数及体重波动对乳腺癌患者上肢淋巴水肿的影响[J]. 中 国 康 复 医 学 杂 志 ,2020,35(2):182-185. D0I:10.3969/j.issn.1001-1242.2020.02.011.
- [4] 赵启超. 下肢十二个穴位浅淋巴管的观察[J]. 中医药学报,2000,(02):56-57.DOI:10.19664/j.cnki.1002-2392.2000.02.055.
- [5] 曾荣华, 欧阳厚淦, 周露, 等. 经络与淋巴系统关系的研究概况 [J]. 中国中医基础医学杂志, 2018, 24(08):1181-1183. DOI:10. 19945/j. cnki. issn. 1006-3250. 2018. 08. 054.
- [6] 颜培宇. 不同穴位针刺对免疫抑制大鼠神经肽相关基因表达及免疫调节作用的分子机制研究 [D]. 黑龙江中医药大学,2010.
- [7] 郭慧娟. 经络按摩联合中药溻渍治疗乳腺癌术后上肢淋巴水肿的临床观察 [J]. 中国民间疗法,2022,30(18):71-73+76. DOI:10. 19621/j. cnki. 11-3555/r. 2022. 1823.
- [8] 方丹萍, 陈亮. 经络按摩联合中医外治法治疗乳腺癌术后淋巴水肿的护理体会 [J]. 中国医药指南, 2017, 15 (14): 270. DOI: 10. 15912/j. cnki. gocm. 2017. 14. 222.